CLINICAL TRIAL: NCT01076361
Title: Medtronic Model 4968 CapSure Epi® Steroid-Eluting Bipolar Epicardial Pacing Lead Post-approval Study
Brief Title: Model 4968 CAPTURE EPI® STERIOD-ELUTING BIPOLAR EPICARDIAL PACING LEAD Post-approval Study
Acronym: 4968
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 4968
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Arrhythmia; Heart Failure
Keywords: Epicardial; Pacing Lead
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The Medtronic CapSure Epi Lead Post-approval Study will assess long-term safety of the 4968 lead. This study is part of the Medtronic System Longevity Study.

DETAILED DESCRIPTION:
The Medtronic CapSure Epi Lead Post-approval Study is being conducted as part of the requirements to satisfy the PMA conditions of approval for the Model 4968 lead. 100 subjects (adult and pediatric) with a 4968 lead will be followed for a minimum of five years to assess the long-term safety of the leads.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent and/or authorization for access to and use of health information by subjects or appropriate legal guardians as required by an institution's Investigational Review Board, Medical Ethics Board, or Research Ethics Board
* Availability of implant, follow-up, and product-related event data
* Implanted with a Model 4968 Capsure Epi Lead

Exclusion Criteria:

* Subjects receiving an implant of a Medtronic lead at a non-participating center and the implant data and current status cannot be confirmed within 30 days after implant
* Subjects who are, or will be inaccessible for follow-up at a 4968 Post-approval study center
* Subjects implanted with a Medtronic cardiac therapy device whose predetermined enrollment limit for that specific product has been exceeded
* Subjects with exclusion criteria required by local law

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects implanted with a 4968 lead.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 1999-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 4968 Clinical Trial Leader, Study Chair — Medtronic
Locations (106):
- United States (83):
  - Alaska Heart Institute, Anchorage, Alaska
  - Gilbert, Arizona
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Bakersville, California
  - Chula Vista, California
  - Downey, California
  - East Palo Alto, California
  - Los Angeles, California
  - Salinas, California
  - Torrance, California
  - Van Nuys, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Ocala, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Marietta, Georgia
  - Oak Lawn, Illinois
  - Indianapolis, Indiana
  - Newburgh, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Alexandria, Louisiana
  - Baton Rouge, Louisiana
  - Salisbury, Maryland
  - Silver Spring, Maryland
  - Towson, Maryland
  - Grand Blanc, Michigan
  - Marquette, Michigan
  - Saginaw, Michigan
  - Southfield, Michigan
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - Lebanon, New Hampshire
  - Browns Mills, New Jersey
  - Newark, New Jersey
  - Ocean City, New Jersey
  - Parlin, New Jersey
  - West Orange, New Jersey
  - Albuquerque, New Mexico
  - Mineola, New York
  - Rochester, New York
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Doylestown, Pennsylvania
  - Lancaster, Pennsylvania
  - Sayre, Pennsylvania
  - Columbia, South Carolina
  - Florence, South Carolina
  - Sioux Falls, South Dakota
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Burlington, Vermont
  - Chesapeake, Virginia
  - Fairfax, Virginia
  - Olympia, Washington
  - Spokane, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Bedford Park, South Australia, Australia
- Austria (2):
  - Linz
  - Vienna
- Hasselt, Belgium
- Canada (7):
  - Calgary, Alberta
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Ste-Foy, Quebec
  - Regina, Saskatchewan
- Copenhagen, Denmark
- Marseille, France
- Homburg/Saar, Germany
- Italy (3):
  - Catanzaro
  - Reggio Emilia
  - Udine
- Netherlands (2):
  - Eindhoven
  - Rotterdam
- Belgrade, Serbia and Montenegro
- Valencia, Spain
- Skövde, Sweden
- Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All enrolled patients with at least 1 Model 4968 lead implanted
Groups:
- Model 4968 Leads: A total of 631 leads were implanted in 370 patients. 22 leads in 21 patients were excluded from analysis.
Period: Overall Study
Arm/Group | Model 4968 Leads
Started | 370 (631 leads were implanted in 370 patients. 22 leads in 21 patients were excluded from analysis.)
Completed | 349 (Follow-up data was not available for 21 participants (22 leads))
Not Completed | 21
Not completed — 22 leads were excluded from analysis | 21

BASELINE CHARACTERISTICS:
Population: A total of 631 leads were implanted in 370 subjects. 22 leads in 21 patients were not included in the analysis due to missing data. The final number of leads analyzed was 609.
Groups:
- All Enrolled Patients: All patients who were enrolled and implanted with a Model 4968 Lead
Arm/Group | All Enrolled Patients
Number analyzed (Participants) | 370
Age, Customized [Number; unit: participants]
  Unknown | 21
  0 - 12 Years | 155
  13 - 19 Years | 49
  20 + Years | 145
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138
  Male | 232
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 5
  Hispanic or Latino | 1
  White | 16
  Race/Ethnicity not collected | 345
  Other | 1
  Not Reportable per Local Laws/Regulations | 2

OUTCOME MEASURES:

1. Primary Outcome: Survival Probability of the Model 4968 Lead Based on Lead-related Complications
Description: The survival analysis takes into account: Enrolled participants, lead follow-up time, and adjudicated lead related complications. The life-table method was used to analyze lead survival probability.
Time Frame: The requirement to satisfy the PMA condition of Approval of model 4968 was to have 100 participants followed for a minimum of 5 years to assess the long-term safety.
Population: 22 Model 4968s (in 21 participants) was not available for analysis
Measure: Number (95% Confidence Interval); unit: percentage of Model 4968 Leads
Units Other Than Participants: leads
Groups:
- Model 4968 Lead Survival Probability: Model 4968 is steroid-eluting bipolar epicardial pacing lead. Participants implanted with Model 4968 lead their data will be obtained for long-term safety and lead events, includes the survival probability for the Model 4968.
Arm/Group | Model 4968 Lead Survival Probability
Number analyzed (Participants) | 349
Number analyzed (leads) | 609
percentage of Model 4968 Leads | 92.3 [88.3 to 95.04]

ADVERSE EVENTS:
Time Frame: Post Implant
Description: All reported lead related events were adjudicated by a technical review committee and reconciled with Medtronic's Event Analysis Reporting System.
Groups:
- Model 4968 Participants: All Model 4968 participants in the analysis cohort
Arm/Group | Model 4968 Participants
Serious Adverse Events (participants affected / at risk) | 30/349
Other Adverse Events (participants affected / at risk) | 0/349
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Model 4968 Participants (N=349)
Over-sensing (Cardiac disorders) | 6 (6)
Insulation breach (Cardiac disorders) | 2 (2)
High impedance (Cardiac disorders) | 3 (3)
Lead conductor fracture (Cardiac disorders) | 6 (6)
Failure to capture/loss of capture (Cardiac disorders) | 13 (13)
Threshold rise, Sudden (Cardiac disorders) | 1 (1)
Failure to sense (Cardiac disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less